CLINICAL TRIAL: NCT05165680
Title: Effect of Aerobic Exercise and Diet on Anthropometric and Hematological Measurements in Obese Anemic Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Nabil Fathy Ahmed, physical therapy practitioner, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003337
Record Dates: First submitted 2021-11-07; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Iron Deficiency Anemia
MeSH Terms: conditions — Obesity; Anemia, Iron-Deficiency | interventions — Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Sixty anemic obese premenopausal women, their ages will range from 30 to 40 years. The participants will be selected from General Zagazig Hospital. All participants will be randomly assigned into two groups equal in number; Experimental group and control group. Experimental group will receive a program of aerobic exercise, low caloric diet rich in iron, vitamin c, and folate for 3 times per week and Iron supplements for 12 weeks , while control group will only receive low caloric diet rich in iron, vitamin c, and folate for 3 times per week and Iron supplements for 12 weeks . Participants' demographic data will be collected as marital status, length of menstrual cycle, level of income, level of education, occupation.
Who Masked: Participant, Investigator
Masking Description: double blinded as neither the subjects nor the investigators are aware of the treatment assignment until the end of the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group, group A (Experimental): Thirty patients in this group will perform aerobic exercise in the form of walking on electric treadmill three times/ week day after day and low caloric diet rich in iron, vitamin C and folate and iron supplement for 12 weeks.
  Interventions: Combination Product: combination of aerobic exercise and healthy diet
- healthy diet (Active Comparator): ow caloric diet rich in iron, vitamin C and folate and iron supplement for 12 weeks.
  Interventions: Combination Product: combination of aerobic exercise and healthy diet

INTERVENTIONS:
Combination Product: combination of aerobic exercise and healthy diet — The 30 patients in this group will receive iron supplements, a personalized low caloric diet therapy based on Harris-Benedict equation. A restricted balanced diet will be prescribed which will be included. Perform aerobic exercise in the form of walking on electrical treadmill three times/ week day after day for 12 weeks according to following parameters.
  * Type: moderate treadmill aerobic exercise
  * Time: 40 minutes (5 minutes warm up phase, 30 minutes target heart rate (THR) phase, 5 minutes cooling down phase)
  * Intensity: THR will be at 75% of maximum heart rate (which will be determined by submaximal graded exercise test and predicated MHR=220-age)
  * Frequency: three times per week for 12 weeks

SUMMARY:
Obesity and iron deficiency (ID) are two forms of the most usual nutritional disorders worldwide. Iron deficiency remains the most common nutritional deficiency and cause of anemia worldwide. Populations in the developing countries, premenopausal females, pregnant women, children, vegetarians and frequent blood donors are largely affected by iron deficiency due to low dietary intake, inadequate bioavailable iron, increased iron demand required for growth and development, iron losses and changes in blood volume. WHO recognized obesity as disease, which is prevalent in both developing and developed countries. Overweight and obesity are now so common and thereby replacing the more traditional public health concerns (under nutrition and infectious diseases) as some of most significant contributors to ill health.

The aim of this study is to investigate effect of aerobic exercise and diet on obese anemic premenopausal women which not clarified previously.

It will be hypothesized that:

There will be no significant effect of aerobic exercise and diet on the anthropometric and hematological measurements in obese anemic women.

DETAILED DESCRIPTION:
Low level of serum iron was observed with weight gain and increasing BMI, both iron deficiency and obesity are worldwide epidemics affecting billions with regional variation.

Iron-deficiency anemia has a substantial effect on the lives of premenopausal women in both low-income and developed countries. A low level of iron, leading to anemia, can result from various causes. The causes of iron-deficiency anemia are pregnancy or childhood growth spurts, Heavy menstrual periods. Iron-deficiency anemia is chronic and frequently asymptomatic and thus may often go undiagnosed. Symptoms include tiredness, lethargy, feeling faint and becoming breathless easily, headaches, irregular heartbeats (palpitations), altered taste, sore mouth and ringing in the ears (tinnitus). Anemia in pregnancy increases the risk of complications in both mother and baby such as low birth weight baby, preterm (premature) delivery and postnatal depression. Low iron reserves in the baby may also lead to anemia in the newborn baby.

Several factors may explain why greater adiposity increases risk for anemia. However, even if diets of overweight individuals are not lower in iron, the absorption of the iron may be reduced because increased circulating hepcidin (a 25-amino-acid peptide hormone with a key role in body iron regulation, is produced mainly by the liver but also, possibly, by adipose tissue in obesity may reduce iron absorption, Iron requirements in overweight individuals may be increased due to larger blood volume and higher basal iron losses with higher body weight. women suggest greater adiposity is associated with lower fractional iron absorption in humans.

Exercise training can increase total Hb and red cell mass, which enhances oxygen-carrying capacity. The possible underlying mechanisms are proposed to come mainly from bone marrow, including stimulated erythropoiesis with hyperplasia of the hematopoietic bone marrow, improvement of the hematopoietic microenvironment induced by exercise training, and hormone- and cytokine-accelerated erythropoiesis. The effects of exercise training on counteracting anemia have been explored and evaluated. The results of the research available to date are controversial, and it seems that significant methodological limitations exist. However, exercise training might be a promising, additional, safe and economical method to help improve anemia. There is a need for further investigation into the effects of and guidelines for exercise interventions in this population of patients.

Largely, the prevailing evidence suggests that a healthy mode of weight loss in obese subjects is accompanied by an improvement of inflammatory markers along with re-established dietary iron absorption and serum iron concentrations as an indication for re-establishment of physiological iron homeostasis. Treating anemia is a matter of how much food we eat that aid in hemoglobin synthesis. In general, to treat anemia, focus should be placed on foods that are good sources of iron, copper, zinc, folic acid, Vitamin B-12, protein, fruits, vegetables, meat, honey, legumes and nuts.

Sixty anemic obese premenopausal women participants, their ages will range from 30 to 40 years. The participants will be selected from General Zagazig Hospital. All participants will be randomly assigned into two groups equal in number; Experimental group and control group. Experimental group will receive a program of aerobic exercise, low caloric diet rich in iron, vitamin c, and folate for 3 times per week and Iron supplements for 12 weeks , while control group will only receive low caloric diet rich in iron, vitamin c, and folate for 3 times per week and Iron supplements for 12 weeks . Participants' demographic data will be collected as marital status, length of menstrual cycle, level of income, level of education, occupation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age will ranges from 30 to 40 years. 2. BMI will ranges from 30 to 34.9 kg/m2 3. Hemoglobin level will ranges from 8 to 11 g/dl. 4. All of participants suffer from iron deficiency anemia. 5. Same level of physical activity according to physical activity index. 6. Same level of education and income.

Exclusion Criteria:

* 1. Cognitive impairment that prevents participants from performing the evaluations and who are unable to understand and sign the written informed consent.

  2. Hypertension. 3. diabetes mellitus 4. Disabling musculoskeletal disorder. 5. Patients with coronary artery disease or heart failure 6. Peripheral vascular disease in lower limb as deep venous thrombosis. 7. Stroke and bone disease, renal, liver, endocrinal disorders, cancer, or chemotherapy.

  8. Different types of anemia. 9. Worms' affection. 10. Pregnancy and lactation. 11. Vitamins deficiency. 12. Six months post large surgeries.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — all participants are married women with normal menstrual cycle
Enrollment: 60 (Estimated)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
BMI in kg/m2 | 3 months
  The anthropometric measurements will be detected via the in body scale. BMI (kg/m2) will be measured for all participants by dividing each participant's body weight (kg) by their heights (m2). Further, WC will be estimated during full expiration using an elastic tape midway between the last rib and the upper iliac crest border.

SECONDARY OUTCOMES:
RBCs in cells/ml | 3 months
  Blood sample analysis to show the hematological measurements level, each participant will be asked to lie in half- lying position, with well supported back and arms. The antecubital area will be cleaned with alcohol. Blood sample will be drawn from the brachial vein from all participants by disposable sterile syringe.
HB in g/dl | 3 months
  blood sample analysis
MCV in fl/cell | 3 months
  blood sample analysis
MCH in pg/cell | 3 months
  blood sample analysis
MCHC in g/dl | 3 months
  blood sample analysis
RDW in % | 3 months
  blood sample analysis
WBCs /mm3 | 3 months
  blood sample analysis
Platelets count /mm3 | 3 months
  blood sample analysis
serum ferritin in ng/ml | 3 months
  blood sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: gehan elmeniawy, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing study protocols with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years after completion
Access Criteria: publishing journal
URL: http://Scholar.cu.edu.eg/p_t